CLINICAL TRIAL: NCT04186845
Title: A Prospective, Phase 3, Multi Center, Single-arm, Imaging Study Investigating the Safety and Diagnostic Performance of rhPSMA 7.3 (18F) PET Ligand in Men With Suspected Prostate Cancer Recurrence Based on Elevated PSA Following Prior Therapy (SPOTLIGHT)
Brief Title: Imaging Study to Investigate Safety and Diagnostic Performance of 18F rhPSMA 7.3 PET Ligand in Suspected Prostate Cancer Recurrence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Blue Earth Diagnostics (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BED-PSMA-302
Record Dates: First submitted 2019-11-22; First posted 2019-12-05 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Recurrent Prostate Cancer; Diagnostic; Prostate Specific Membrane Antigen (PSMA); Positron Emission Tomography (PET) Scan
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Injections; Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: Positron Emission Tomography (PET) Imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  Interventions: Drug: rhPSMA-7.3 (18F) Injection; Diagnostic Test: Positron emission tomography scan

INTERVENTIONS:
Drug: rhPSMA-7.3 (18F) Injection — Radioligand for PET CT scanning
  Other Names: flotufolastat F18
Diagnostic Test: Positron emission tomography scan — Imaging scan with radioligand
  Other Names: PET scan

SUMMARY:
A prospective, Phase 3, multi center, single-arm, imaging study investigating the safety and diagnostic performance of rhPSMA 7.3 (18F) Positron Emission Tomography (PET) ligand in men with suspected prostate cancer recurrence based on elevated Prostate-specific antigen (PSA) following prior therapy.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the patient-level correct detection rate (CDR) and region-level positive predictive value (PPV) of rhPSMA-7.3 (18F) positron emission tomography (PET) for biochemical recurrence (BCR) of prostate cancer using histopathology or imaging as a standard of truth (SoT).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male and aged >18 years old.
2. History of localized adenocarcinoma of the prostate with prior curative intent treatment.
3. An elevated PSA, clinically suspicious for biochemically recurrent disease:

   * Following Radical Prostatectomy: PSA >0.2 ng/mL
   * Following Radiotherapy: nadir +2 ng/mL.
4. Potentially eligible for salvage therapy with curative intent.

Exclusion Criteria:

1. Patients who are planned to have an x-ray contrast agent or other PET radiotracer <24 hours prior to the PET scan.
2. Patients currently receiving Androgen Deprivation Therapy (ADT).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients required to have suspected prostate cancer recurrence based on elevated PSA following prior therapy.
Enrollment: 391 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Tower Urology, Los Angeles, California
  - University of California Irvine Medical Center (UCIMC), Orange, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Austell, Georgia
  - Northshore University HealthSystem, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - University of Michigan Ann Arbor, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Queens Hospital Center (QHC - Queens Cancer Center, Jamaica, New York
  - Mount Sinai Faculty Practice Associates, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Hospital, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - MidLantic Urology, Philadelphia, Pennsylvania
  - MD Anderson Hospital, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - University of Virginia - Health Science Center, Charlottesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Turku University Hospital, Turku, Finland
- Netherlands (2):
  - CWZ, Nijmegen
  - Maxima MC, Veldhoven

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 04 May 20 (first patient, screening visit) and 12 Oct 21 (database lock), with last patient, last visit on 28 Apr 21. It was conducted at 28 activated study sites (27 recruited) in 3 countries. Of the 420 patients screened, 391 patients met all the study eligibility criteria
Pre-assignment Details: Baseline safety evaluations performed at screening (Visit 1) comprised vital signs and recording of any adverse events (AEs) from the time of informed consent. Conventional images collected within 90 days of rhPSMA7.3 (18F) PET, followed by biopsy within 60 days post-PET scan or confirmatory imaging within 90 days post-PET scan
Groups:
- Single Arm: All patients who were scheduled to receive the rhPSMA-7.3 (18F) injection having met the inclusion/exclusion criteria or who received the rhPSMA-7.3 (18F) injection.
Period: Overall Study
Arm/Group | Single Arm
Started | 391
Completed | 378
Not Completed | 13
Not completed — Death | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Biopsy ordered but area too small to biopsy | 1
Not completed — Biopsy ordered but not done | 1
Not completed — It was previously confirmed | 1
Not completed — Patient cancelled scheduled scans | 2
Not completed — PSMA PET/CT scan show disease within previously Bx area | 1
Not completed — Subject refused confirmatory imaging | 1
Not completed — Too small to biopsy | 1

BASELINE CHARACTERISTICS:
Population: All patients who were scheduled to receive the rhPSMA-7.3 (18F) injection having met the inclusion/exclusion criteria or who received the rhPSMA-7.3 (18F) injection.
Groups:
- Single Arm: Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  rhPSMA-7.3 (18F) Injection: Radioligand for PET CT scanning
  Positron emission tomography scan: Imaging scan with radioligand
Arm/Group | Single Arm
Number analyzed (Participants) | 391
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 121
  >=65 years | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 391
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 342
  Unknown or Not Reported | 31
Race/Ethnicity, Customized [Number; unit: participants] — Race split into 3 substantive categories and also those for whom it was not reported
  participants
    Black or African American | 61
    White | 295
    Other | 14
    Not Reported | 21
Region of Enrollment [Number; unit: participants]
  Netherlands | 9
  United States | 375
  Finland | 7
Total Gleason Score [Number; unit: participants] — Gleason score (defined by the International Society of Urological Pathologists) was based on prostate biopsy.
  Score 6 - The cells look similar to normal prostate cells. The cancer is likely to grow very slowly, if at all
  Score 7 - Most cells still look similar to normal prostate cells. The cancer is likely to grow slowly
  Score 8 - Some cells look abnormal. The cancer might grow quickly or at a moderate rate
  Score 9 or 10 - The cells look very abnormal. The cancer is likely to grow quickly
  participants
    ≤6 | 39
    =7 | 232
    =8 | 41
    =9 | 63
    =10 | 1
    Missing | 15
Gleason Grade Group (GGG) [Number; unit: participants] — GGG (defined by the International Society of Urological Pathologists) was based on prostate biopsy.
  Group 1: The cells look similar to normal prostate cells. The cancer is likely to grow very slowly, if at all
  Group 2: Most cells still look similar to normal prostate cells. The cancer is likely to grow slowly
  Group 3: The cells look less like normal prostate cells. The cancer is likely to grow at a moderate rate
  Group 4: Some cells look abnormal. The cancer might grow quickly or at a moderate rate
  Group 5: The cells look very abnormal. The cancer is likely to grow quickly
  participants
    =1 | 39
    =2 | 104
    =3 | 116
    =4 | 41
    =5 | 64
    Missing | 27
TNM (Tumor-Node-Metastasis) Stage T [Number; unit: participants] — Pathological TNM stage was used if available, otherwise the clinical TNM was used.
  T1 means the cancer is too small to be seen on a scan, or felt during an examination of the prostate T1a means that the cancer is in less than 5% of the removed tissue T1c cancers are found by biopsy T2 means the cancer is completely inside the prostate gland T3a means the cancer has broken through the capsule (covering) of the prostate gland T3b means the cancer has spread into the tubes that carry semen (seminal vesicles) T4 means the cancer has spread into other body organs nearby
  participants
    T1 | 4
    T1c | 54
    T2 | 52
    T2a | 15
    T2b | 10
    T2c | 63
    T3 | 10
    T3a | 82
    T3b | 68
    T4 | 2
    TX | 7
    Missing | 24
TNM Stage N [Number; unit: participants] — Pathological TNM stage was used if available, otherwise the clinical TNM was used.
  N0 means that the nearby lymph nodes don't contain cancer cells
  N1 means there are cancer cells in lymph nodes near the prostate
  participants
    N0 | 249
    N1 | 53
    NX | 61
    Missing | 28
TNM Stage M [Number; unit: participants] — Pathological TNM stage was used if available, otherwise the clinical TNM was used.
  M0 means the cancer hasn't spread to other parts of your body.
  M1 means the cancer has spread to other parts of the body outside the pelvis. It is split into M1a, M1b and M1c.
  M1a means there are cancer cells in lymph nodes outside the pelvis
  M1b means there are cancer cells in the bone
  M1c means there are cancer cells in other parts of the body such as the lungs
  participants
    M0 | 243
    M1 | 1
    M1b | 1
    MX | 106
    Missing | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] — BMI was calculated as weight in kg divided by height in m2. Population: Not all subjects had height and weight measured (eg only 337 subjects had height at baseline) - the trial was conducted during the Covid pandemic.
  Kg/m2
    number analyzed (Participants) | 334
    (all) | 28.68 (4.740)
Time since initial cancer diagnosis [Mean (Standard Deviation); unit: months] — Population: Date of cancer diagnosis was not available for 2 participants.
  months
    number analyzed (Participants) | 389
    (all) | 87.3 (65.70)
Time since diagnosis of biochemical recurrence [Mean (Standard Deviation); unit: months] — Population: Date of diagnosis of biochemical recurrence not available for all participants
  months
    number analyzed (Participants) | 390
    (all) | 17.1 (27.15)
Time since start of adjuvant treatment [Mean (Standard Deviation); unit: months] — Population: Not all participants had adjuvant treatment and start date not always available for all participants who had adjuvant treatment.
  months
    number analyzed (Participants) | 190
    (all) | 67.3 (50.26)
Time since end of adjuvant treatment [Mean (Standard Deviation); unit: months] — Population: Not all participants had adjuvant treatment and end date not always available for all participants who had adjuvant treatment.
  months
    number analyzed (Participants) | 192
    (all) | 60.2 (49.11)
Duration of adjuvant treatment [Mean (Standard Deviation); unit: months] — Population: Not all participants had adjuvant treatment and start and end dates not always available for all participants who had adjuvant treatment in order to calculate duration.
  months
    number analyzed (Participants) | 187
    (all) | 7.2 (16.05)

OUTCOME MEASURES:

1. Primary Outcome: Patient-level CDR and Region-level PPV of rhPSMA7.3 (18F) PET for BCR of Prostate Cancer Using Histopathology or Imaging as a SoT
Description: The CDR was defined as the percentage of all patients scanned who had at least one TP lesion (localized correspondence between rhPSMA-7.3 (18F) PET imaging and the reference standard) regardless of any coexisting FP findings. When determining the region-level PPV, all rhPSMA7.3 (18F) PET-positive regions (maximum of three per patient) were categorized as TP or FP regions using histopathology or imaging.
Time Frame: Conventional images within 90 days of rhPSMA7.3 (18F) PET, followed by biopsy within 60 days post-PET scan or confirmatory imaging within 90 days post-PET scan
Population: Patients who received rhPSMA-7.3 (18F) injection followed by a PET/CT scan and for whom sufficient data are available to permit a clear classification following the SoT algorithm.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Efficacy Analysis Population (EAP): Patients who received rhPSMA-7.3 (18F) injection followed by a PET/CT scan and for whom sufficient data are available to permit a clear classification following the SoT algorithm.
Arm/Group | Efficacy Analysis Population (EAP)
Number analyzed (Participants) | 366
percentage
  Patient-level CDR - Central Reader 1 | 54.1 [48.8 to 59.3]
  Patient-level CDR - Central Reader 2 | 51.4 [46.1 to 56.6]
  Patient-level CDR - Central Reader 3 | 51.6 [46.4 to 56.9]
  Region-level PPV - Central Reader 1 | 46.2 [42.0 to 50.3]
  Region-level PPV - Central Reader 2 | 60.3 [55.1 to 65.5]
  Region-level PPV - Central Reader 3 | 52.6 [47.6 to 57.5]

2. Secondary Outcome: Patient-level CDR and Region-level PPV of rhPSMA-7.3 (18F) PET in Patients Who Had Negative Baseline Conventional Imaging
Description: Patient-level CDR was defined as the percentage of all patients scanned who had at least one TP lesion (localized correspondence between rhPSMA-7.3 (18F) PET imaging and the reference standard) regardless of any co-existing FP findings.
  Region-Level PPV is defined as the regions which are true positive out of all regions with positive lesions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Efficacy Analysis Population (EAP)
Number analyzed (Participants) | 250
percentage
  Patient Level CDR - Central Reader 1 | 46.8 [40.5 to 53.2]
  Patient Level CDR - Central Reader 2 | 45.2 [38.9 to 51.6]
  Patient Level CDR - Central Reader 3 | 45.6 [39.3 to 52.0]
  Region-level PPV - Central Reader 1 | 39.7 [34.6 to 44.9]
  Region-level PPV - Central Reader 2 | 56.2 [49.6 to 62.7]
  Region-level PPV - Central Reader 3 | 46.8 [40.7 to 52.9]

3. Secondary Outcome: Patient-level CDR and Region-level PPV of rhPSMA-7.3 (18F) PET for Recurrence in Those Patients With and Without Reference Standard Histopathology Available
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Efficacy Analysis Population (EAP): all patients who received rhPSMA-7.3 (18F) injection followed by a PET/CT scan and for whom sufficient data are available to permit a clear classification following the SoT algorithm.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Histopathology Available as SoT: Patients with Histopathology available as SoT
- Histopathology Not Available as SoT: Patients without histopathology available as SoT
Arm/Group | Histopathology Available as SoT | Histopathology Not Available as SoT
Number analyzed (Participants) | 69 | 297
percentage
  Patient-level CDR - Central Reader 1 | 75.4 [63.5 to 84.9] | 49.2 [43.3 to 55.0]
  Patient-level CDR - Central Reader 2 | 76.8 [65.1 to 86.1] | 45.5 [39.7 to 51.3]
  Patient-level CDR - Central Reader 3 | 73.9 [61.9 to 89.7] | 46.5 [40.7 to 52.3]
  Region-level PPV - Central Reader 1 | 60.9 [52.0 to 69.8] | 42.4 [37.7 to 47.0]
  Region-level PPV - Central Reader 2 | 67.0 [57.6 to 76.4] | 57.9 [51.7 to 64.0]
  Region-level PPV - Central Reader 3 | 62.6 [53.5 to 71.8] | 49.5 [43.8 to 55.3]

4. Secondary Outcome: Patient-level CDR of rhPSMA-7.3 (18F) PET Stratified by PSA Level
Description: Patient-level CDR was defined as the percentage of all patients scanned who had at least one TP lesion (localized correspondence between rhPSMA-7.3 (18F) PET imaging and the reference standard) regardless of any co-existing FP findings. The last PSA level before the PET scan will be used to stratify the patients
Time Frame: as for outcome 1
Population: Efficacy Analysis Population (EAP): all patients who received rhPSMA-7.3 (18F) injection followed by a PET/CT scan and for whom sufficient data are available to permit a clear classification following the SoT algorithm, and with baseline PSA available
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- PSA<0.5: PSA < 0.5
- 0.5≤PSA<1.0: 0.5 ≤ PSA < 1.0
- 1.0≤PSA<2.0: 1.0 ≤ PSA < 2.0
- 2.0≤PSA<5.0: 2.0 ≤ PSA < 5.0
- 5.0≤PSA<10.0: 5.0 ≤ PSA < 10.0
- PSA≥10.0: PSA ≥ 10.0
Arm/Group | PSA<0.5 | 0.5≤PSA<1.0 | 1.0≤PSA<2.0 | 2.0≤PSA<5.0 | 5.0≤PSA<10.0 | PSA≥10.0
Number analyzed (Participants) | 105 | 63 | 43 | 88 | 36 | 31
percentage
  Central Reader 1 | 29.5 [21.0 to 39.2] | 44.4 [31.9 to 57.5] | 65.1 [49.1 to 79.0] | 72.7 [62.2 to 81.7] | 61.1 [43.5 to 76.9] | 80.7 [62.5 to 92.5]
  Central Reader 2 | 23.8 [16.0 to 33.1] | 41.3 [29.0 to 54.4] | 65.1 [49.1 to 79.0] | 70.5 [59.8 to 79.7] | 58.3 [40.8 to 74.5] | 83.9 [66.3 to 94.5]
  Central Reader 3 | 25.7 [17.7 to 35.2] | 46.0 [33.4 to 59.1] | 62.8 [46.7 to 77.0] | 69.3 [58.6 to 78.7] | 58.3 [40.8 to 74.5] | 77.4 [58.9 to 90.4]

5. Secondary Outcome: CDR of rhPSMA-7.3 (18F) PET in the Following Regions: Prostate/Prostate Bed, Pelvic Lymph Nodes, Other
Description: Patient-level CDR was defined as the percentage of all patients scanned who had at least one TP lesion (localized correspondence between rhPSMA-7.3 (18F) PET imaging and the reference standard) regardless of any co-existing FP findings. The analysis was performed for each region and for each of the blinded independent readers
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Prostate/ Prostate Bed: Prostate or prostate bed
- Pelvic Lymph Nodes: Pelvic Lymph Nodes
- Other (Extra-pelvic) Sites: Other (extra-pelvic) sites
Arm/Group | Prostate/ Prostate Bed | Pelvic Lymph Nodes | Other (Extra-pelvic) Sites
Number analyzed (Participants) | 366 | 366 | 366
percentage
  Central Reader 1 | 16.7 [13.0 to 20.9] | 21.6 [17.5 to 26.2] | 29.2 [24.6 to 34.2]
  Central Reader 2 | 13.1 [9.8 to 17.0] | 19.4 [15.5 to 23.8] | 30.6 [25.9 to 35.6]
  Central Reader 3 | 13.7 [10.3 to 17.6] | 22.4 [18.2 to 27.0] | 25.7 [21.3 to 30.5]

6. Secondary Outcome: Percentage of Patients in Whom rhPSMA-7.3 (18F) PET Imaging Results Changed the Intended Patient Management (Major and Other Changes)
Description: This analysis used patients in the EAP who had documented patient management plans in the EDC before and after the rhPSMA-7.3 (18F) PET scan
Time Frame: as for outcome 1
Population: Patients in the EAP who had documented patient management plans in the EDC before and after the rhPSMA-7.3 (18F) PET scan.
Measure: Number; unit: percentage
Groups:
- Change in Management Plan: Change in Management Plan for patients with both pre-PSMA and post-PSMA management plans
Arm/Group | Change in Management Plan
Number analyzed (Participants) | 167
percentage
  No Change | 6.6
  Major Change | 46.7
  Minor Change | 4.8
  Additional Information Required | 31.7
  Pre-PSMA Plan Not Valid | 10.2

7. Secondary Outcome: Reader Kappa Statistics of rhPSMA7.3 (18F) Scan Interpretation by the Blinded Independent Readers
Description: The Cohen's kappa statistic will be calculated to assess pairwise agreement between any 2 blinded independent readers
Time Frame: PET Scan on Day 1
Population: Evaluable PET Scan Population (EPSP): All patients who received the rhPSMA-7.3 (18F) injection with a PET scan.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Patient-level Inter-reader Reproducibility: Patient-level Inter-reader Reproducibility for Evaluable PET Scan Population (EPSP)
Arm/Group | Patient-level Inter-reader Reproducibility
Number analyzed (Participants) | 389
percentage
  Central Reader 1 vs Reader 2 | 0.29 [0.21 to 0.38]
  Central Reader 1 vs Reader 3 | 0.38 [0.25 to 0.51]
  Central Reader 2 vs Reader 3 | 0.50 [0.41 to 0.60]

8. Secondary Outcome: Region-level PPV of rhPSMA-7.3 (18F) PET Stratified by PSA Level
Description: Region-Level PPV is defined as the regions which are true positive out of all regions with positive lesions.. The last PSA level before the rhPSMA-7.3 (18F) PET scan was used to stratify patients.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- PSA <0.5: PSA < 0.5
Arm/Group | PSA <0.5 | 0.5≤PSA<1.0 | 1.0≤PSA<2.0 | 2.0≤PSA<5.0 | 5.0≤PSA<10.0 | PSA≥10.0
Number analyzed (Participants) | 105 | 63 | 43 | 88 | 36 | 31
percentage
  Central Reader 1 | 29.1 [20.5 to 37.7] | 37.1 [27.6 to 46.6] | 45.6 [35.1 to 56.1] | 57.7 [50.1 to 65.3] | 57.9 [44.9 to 70.9] | 59.6 [47.6 to 71.7]
  Central Reader 2 | 50.8 [36.9 to 64.8] | 51.8 [38.9 to 64.6] | 57.4 [43.7 to 71.1] | 65.0 [55.3 to 74.6] | 71.7 [56.8 to 86.7] | 62.7 [50.6 to 74.9]
  Central Reader 3 | 34.5 [24.0 to 45.0] | 45.1 [33.5 to 56.7] | 52.5 [38.7 to 66.2] | 64.9 [55.9 to 73.9] | 58.7 [41.5 to 75.9] | 60.8 [47.3 to 74.2]

9. Secondary Outcome: Region-level PPV of rhPSMA-7.3 (18F) PET for Recurrence in Those Patients With and Without Reference Standard Histopathology Available
Description: Region-Level PPV is defined as the regions which are true positive out of all regions with positive lesions. The data are analysed by whether the patients have had histopathology as reference standard.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Histopathology Available as SoT; Histopathology Not Available as SoT: Region-level PPV, Region-level 95% CIs were calculated via clustered binary data algorithm.
Arm/Group | Histopathology Available as SoT | Histopathology Not Available as SoT
Number analyzed (Participants) | 69 | 297
percentage
  Central Reader 1 | 60.9 [52.0 to 69.8] | 42.4 [37.7 to 47.0]
  Central Reader 2 | 67.0 [57.6 to 76.4] | 57.9 [51.7 to 64.0]
  Central Reader 3 | 62.6 [53.5 to 71.8] | 49.5 [43.8 to 55.3]

ADVERSE EVENTS:
Time Frame: AEs were also monitored throughout the study through study completion, an average of 90 days post-IMP administration.
Description: AEs (treatment emergent) were coded with MedDRA and data listed by patient: study site, patient identifier, age, race, AE (MedDRA SOC, PT and verbatim term), dates of onset and resolution, duration, CTCAE toxicity grade, seriousness, action taken, outcome and causality. Deaths, SAEs and AEs leading to discontinuation were listed by patient
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 2/391
Serious Adverse Events (participants affected / at risk) | 2/391
Other Adverse Events (participants affected / at risk) | 28/391
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=391)
Sudden death (General disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=391)
Hypertension (Vascular disorders) | 7 (7)
Flushing (Vascular disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (2)
Injection site discomfort (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT04186845/Prot_003.pdf
  • Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT04186845/SAP_002.pdf